CLINICAL TRIAL: NCT07308132
Title: A Phase 1, First-in-Human Study of a Novel CD79bxCD20xCD3 Trispecific Antibody in B-Cell Non-Hodgkin Lymphoid Malignancies (NHLs)
Brief Title: A Study of JNJ-95566692 in Participants With Non-Hodgkin Lymphoid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 95566692LYM1001; 2025-523297-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: JNJ-95566692 (Experimental): Participants will receive escalating doses of JNJ-95566692 in Part 1 (Dose escalation) to determine the putative recommended Phase 2 doses (RP2D[s]) and dosing schedule(s). Participants in Part 2 (Dose expansion) will receive JNJ-95566692 at the putative RP2D(s) determined in Part 1 to further characterize safety, PK (pharmacokinetic), pharmacodynamic (PD) and clinical activity.
  Interventions: Drug: JNJ-95566692
- Arm B: JNJ-95566692 in combination with JNJ-87801493 (Experimental): Participants will receive escalating doses of JNJ-95566692 in combination with JNJ-87801493 in Part 1 (Dose escalation) to determine the putative RP2D[s] and dosing schedule(s). Participants in Part 2 (Dose expansion) will receive JNJ-95566692 in combination with JNJ-87801493 at the putative RP2D(s) determined in Part 1 to further characterize safety, PK, PD and clinical activity.
  Interventions: Drug: JNJ-95566692; Drug: JNJ-87801493

INTERVENTIONS:
Drug: JNJ-95566692 — JNJ-95566692 will be administered subcutaneously.
Drug: JNJ-87801493 — JNJ-87801493 will be administered subcutaneously.
  Arms: Arm B: JNJ-95566692 in combination with JNJ-87801493

SUMMARY:
The purpose of this study is to determine the putative recommended Phase 2 doses (RP2Ds) and optimal dose schedule(s) for JNJ-95566692 as a single agent (Arm A) and in combination with JNJ-87801493 (Arm B) (Part 1: Dose Escalation) and to further characterize the safety and clinical activity of JNJ-95566692 as a single agent (Arm A) and in combination with JNJ-87801493 (Arm B) at the putative RP2D(s) (Part 2: Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* B-cell non-Hodgkin lymphoid malignancies (NHL) according to World Health Organization (WHO) 2022 with relapsed or refractory disease and no other approved therapies available that would be more appropriate in the investigator's judgment. • Participants must have received at least 2 prior lines of therapy including an αCD20 monoclonal antibody containing chemotherapy combination schedule. • Participants who have received at least one prior line of therapy but are not eligible or do not have access to standard second line therapies, such as CAR-T, will be allowed to enroll
* While on study treatment and for 3 months after the last dose of study treatment, a participant must: not breastfeed or become pregnant; not donate gametes (that is, eggs or sperm) or freeze for future use for the purposes of assisted reproduction; and wear an external condom
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participants must have measurable disease as defined by the disease criteria (Lugano criteria)
* Participants of childbearing potential must have a negative highly sensitive (for example, beta [β]-human chorionic gonadotropin) pregnancy test at screening and within 24 hours before the first dose of study treatment and agree to further pregnancy tests

Exclusion Criteria:

* Known active central nervous system involvement (CNS) or leptomeningeal involvement
* Prior solid-organ transplantation
* Malignancy diagnosis other than the disease under study within 1 year prior to the first dose of the study treatment; exceptions are squamous and basal cell carcinoma of the skin, carcinoma in situ of the cervix and any malignancy that is considered cured or has minimal risk of recurrence within 1 year of first dose of the study treatment in the opinion of both the investigator and sponsor's medical monitor
* Autoimmune or inflammatory disease requiring systemic steroids or other immunosuppressive agents (for example, methotrexate or tacrolimus) within 3 months prior to first dose of study treatment
* Toxicity from prior anticancer therapy that has not resolved to baseline levels or to Grade less than or equal to (<=) 1 (except alopecia, vitiligo, peripheral neuropathy, or Grade <=2 endocrinopathies that are stable on hormone replacement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) by Severity for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  An AE is any untoward medical occurrence in a clinical study participant administered an investigational or non-investigational product and it does not necessarily have a causal relationship with the investigational product. Severity for AEs will be specified as per: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grades which are Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (potentially life-threatening) and Grade 5 (death related to adverse event). SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Part 1: Number of Participants with Dose Limiting Toxicity (DLTs) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Number of participants with DLTs for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported. The DLTs are drug-related toxicities and are defined as any of the following: fatal toxicity, high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Serum Concentration for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Serum concentration for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be assessed using a validated assay method.
Area Under the Curve During a Dosing Interval (AUCtau) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  AUC tau is defined as area under the serum concentration-time curve during a dosing interval (tau).
Maximum Serum Concentration (Cmax) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Cmax for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported.
Minimum Serum Concentration (Cmin) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Cmin for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported.
Area Under the Curve (AUC[0-t]) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  AUC(0-t) for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported.
Half-life (t1/2) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Half-life (t1/2) for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported.
Time to Reach Cmax (Tmax) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Tmax is the time to reach maximum observed serum concentration for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B).
Apparent Total Body Clearance (CL/F) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  CL/F for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported.
Apparent Volume of Distribution (V/F) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  V/F for JNJ-95566692 (arm A) and in combination with JNJ-87801493 (arm B) will be reported.
Number of Participants with Anti-JNJ-95566692 Antibodies in Arm A and Arm B | Approximately 2 years and 8 months
  Participants with presence of antibodies binding to JNJ-95566692 in arm A and arm B will be reported.
Number of Participants with Anti-JNJ-87801493 Antibodies in Arm B | Approximately 2 years and 8 months
  Participants with presence of antibodies binding to JNJ-87801493 in arm B will be reported.
Part 2: Overall Response for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Overall response is defined as a best response of partial response (PR) or better as assessed by the investigator according to standard response criteria per Lugano.
Part 2: Complete Response (CR) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  Complete response (CR) is defined as a best response of CR as assessed by the investigator according to standard response criteria per Lugano.
Part 2: Time to Response (TTR) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  TTR is defined for participants who achieved a response of PR or better as the time from the first dose of study treatment to the first response of PR or better.
Part 2: Duration of Response (DOR) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  DOR is defined for participants who achieved a response of PR or better as the time between the date of initial documentation of first response of PR or better to the date of first documented evidence of progressive disease, initiation of a new systemic anti-cancer therapy or death.
Part 2: Progression-free survival (PFS) for JNJ-95566692 (Arm A) And in Combination With JNJ-87801493 (Arm B) | Approximately 2 years and 8 months
  PFS is defined as the time from the date of first dose of study treatment to the date of first documented evidence of progressive disease (as defined in the disease-specific response criteria; unless) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne
  - Scientia Clinical Research, Randwick
- Turkey (Türkiye) (2):
  - Ankara University Medical Faculty, Ankara
  - Koc University Medical Faculty, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency